CLINICAL TRIAL: NCT03924414
Title: TOPAZ: Trial of Parkinson's And Zoledronic Acid A Randomized Placebo-controlled Trial of Zoledronic Acid for the Prevention of Fractures in Patients With Parkinson's Disease
Brief Title: Trial of Parkinson's And Zoledronic Acid
Acronym: TOPAZ
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of California, San Francisco (Other); Duke University (Other); University of Pittsburgh (Other); Parkinson's Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20180456; 1R01AG059417-01A1 (NIH)
Record Dates: First submitted 2019-04-02; First posted 2019-04-23 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease; Osteoporosis; Parkinsonism; Parkinson's Disease and Parkinsonism; Atypical Parkinsonism; Progressive Supranuclear Palsy; Multiple System Atrophy; Vascular Parkinsonism; Dementia With Lewy Bodies
Keywords: Parkinson Disease; Parkinson's Disease; Osteoporosis; Zoledronic acid; Neurology; Bone; Fracture; Parkinsonism; Atypical Parkinsonism; Progressive Supranuclear Palsy; Multiple System Atrophy; Vascular Parkinsonism; Dementia with Lewy Bodies
MeSH Terms: conditions — Parkinson Disease; Osteoporosis; Parkinsonian Disorders; Supranuclear Palsy, Progressive; Multiple System Atrophy; Lewy Body Disease; Fractures, Bone | interventions — Zoledronic Acid

STUDY DESIGN:
Intervention Model Description: This study is a randomized (1:1) placebo-controlled trial of a single infusion of zoledronic acid-5 mg (ZA) for the prevention of fractures in men and women aged 60 years and older with Parkinson's Disease or parkinsonism with at least 2 years of follow-up.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zoledronic acid (ZA) (Active Comparator): A single intravenous infusion of Zoledronic acid (5 mg) infused over 45 minutes
  Interventions: Drug: Zoledronic Acid 5Mg/Bag 100Ml Inj
- Placebo (Placebo Comparator): A single intravenous infusion of placebo infused over 45 minutes
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Zoledronic Acid 5Mg/Bag 100Ml Inj — Zoledronic acid 5mg/100 ml IV infusion: Zoledronic acid-5 mg (ZA) is an FDA approved therapy for men and postmenopausal women for the treatment and prevention of osteoporosis.
  Other Names: Reclast
  Arms: Zoledronic acid (ZA)
Other: Placebo — Normal Saline 100 ml (placebo) IV infusion
  Arms: Placebo

SUMMARY:
This home-based study is a randomized (1:1) placebo-controlled trial of a single infusion of zoledronic acid-5 mg (ZA) for the prevention of fractures in men and women aged 60 years and older with Parkinson's disease and parkinsonism with at least 2 years of follow-up. A total of 2650 participants will be enrolled and randomized in the United States. Participants, follow-up outcome assessors, and study investigators will be blinded to assigned study treatment. This trial is funded by the National Institute of Aging.

DETAILED DESCRIPTION:
This home-based randomized clinical trial is designed to test the efficacy of ZA-5 mg in Parkinson's disease (PD) and parkinsonism patients. This trial will also address barriers to treatment of patients with PD and parkinsonism by providing rigorous evidence about whether ZA reduces fracture risk in patients with PD and parkinsonism, simplifying treatment by giving ZA at home without extra medical visits and BMD testing, and overcoming poor persistence with oral therapies because one infusion may prevent bone loss for at least 2 years. The outcome of this trial will demonstrate how a home-based fracture prevention can reach older PD patients who would not otherwise receive treatment to reduce their high risk of fractures.

Patients with PD will be recruited throughout the US by participating neurologists and health networks as well as the Parkinson's Foundation. Patients may also self-refer to the study. Interested patients can access study information on a study website (topaz.eurekaplatform.org) as well as through the Parkinson's Foundation Helpline. Patients who wish to enroll will be directed to an interactive electronic consent (eConsent). Following eConsent, participants complete a screening questionnaire (to confirm eligibility), followed by a baseline questionnaire. If a participant is determined to be eligible following these steps, they may be scheduled for a Telemedicine assessment to further confirm the PD or parkinsonism diagnosis, unless they have been referred directly from a participating neurologist. If confirmed, the participant will be mailed a supply of vitamin D3 800-1000 IU and instructed to take one vitamin D tablet every day for 2 months. Lastly, a Nurse Home Visit will be scheduled and conducted to confirm final eligibility, randomization, and administration of the study drug, if appropriate. Participants who are randomized will be contacted every 4 months for at least 2 years to determine if they have had any fractures.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 60 years or older
* Current Parkinson's Disease diagnosis or neurodegenerative parkinsonism diagnosis (including progressive supranuclear palsy, multiple system atrophy, cortical basal degeneration, vascular parkinsonism, dementia with Lewy bodies or another form of neurodegenerative parkinsonism) based on an expert assessment (neurologist diagnosis via medical records confirmation or Telemedicine Screening Assessment)
* Willing and able to continue in follow-up for at least 2 years
* Willing and able to provide informed consent

Exclusion Criteria:

* History of hip fracture
* Any use of a bisphosphonate drug within the last 12 months
* Use of any other osteoporosis treatment (such as SERMs and denosumab) within the last 6 months
* Tooth extraction or invasive dental procedures within the past 30 days or planned/scheduled extraction/procedure in the next 12 months
* Non-ambulatory, i.e., unable to walk without assistance of another person.
* Undergoing kidney dialysis
* A diagnosis of multiple myeloma or Paget's disease
* Unable to speak or read English sufficiently to complete informed consent
* Any other criteria, which would make the patient unsuitable to participate in this study as determined by the study staff (e.g., an uncontrolled drug and/or alcohol addiction)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2650 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Clinical Fractures | 2 years
  All clinical fractures
Number of Participants with Clinical Fractures | 5 years
  All clinical fractures

SECONDARY OUTCOMES:
Number of Participants Hip Fractures | 2 years
  Hip fractures
Number of Participants Hip Fractures | 5 years
  Hip fractures
Mortality | 2 years
  All-cause mortality
Mortality | 5 years
  All-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Steve Cummings, MD, Principal Investigator — CPMC Research Institute
Locations (76):
- United States (76):
  - Mayo Clinic, Scottsdale, Arizona
  - Washington Regional Medical Center, Fayetteville, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sutter Health, Berkeley, California
  - Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - University of California, Irvine, Irvine, California
  - Loma Linda University, Loma Linda, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Valley Parkinson Clinic, Los Gatos, California
  - Parkinson's Disease and Movement Disorder Center of Silicon Valley, Palo Alto, California
  - University of California, Riverside, Riverside, California
  - Sutter Health, Sacramento, California
  - University of California, Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Denver, Aurora, Colorado
  - St. Mary's Medical Center, Grand Junction, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Hartford Healthcare, Hartford, Connecticut
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Parkinson's Foundation, Miami, Florida
  - University of Miami, Miami, Florida
  - Morehouse School of Medicine, Atlanta, Georgia
  - Emory University School of Medicine, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Queens Medical Center, Honolulu, Hawaii
  - Northwestern Medicine, Chicago, Illinois
  - Cook County Health & Hospitals System, Chicago, Illinois
  - Rush University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Loyola University, Chicago, Illinois
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Health System, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Boston University, Boston, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - Quest Research Institute, Farmington Hills, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical College, Albany, New York
  - Stony Brook University Medical Center, East Setauket, New York
  - Northwell Health, Glen Cove, New York
  - Northwell Health, Great Neck, New York
  - Northwell Health, Manhasset, New York
  - New York University Langone Health, New York, New York
  - Mount Sinai Beth Israel, New York, New York
  - Columbia University, New York, New York
  - Weill Cornell Medicine, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Duke University, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, UH Cleveland, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Veracity Neuroscience LLC, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Neurological Institute, Houston, Texas
  - University of Texas Health Houston Medical Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
  - Booth Gardner Parkinson's Care Center at EvergreenHealth, Kirkland, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tanner CM, Cummings SR, Schwarzschild MA, Brown EG, Dorsey ER, Espay AJ, Galifianakis NB, Goldman SM, Litvan I, Luthra N, McFarland NR, Mitchell KT, Standaert DG, Bauer DC, Greenspan SL, Beck JC, Lyles KW. The TOPAZ study: a home-based trial of zoledronic acid to prevent fractures in neurodegenerative parkinsonism. NPJ Parkinsons Dis. 2021 Mar 1;7(1):16. doi: 10.1038/s41531-021-00162-1. PMID 33649343